CLINICAL TRIAL: NCT07385300
Title: Evaluation of the Use of Omega-3 Pufa and Aspirin as Adjunctive Therapy in the Treatment of Smoker Patients With Stage Iii Periodontitis (Randomized Clinical Trial)
Brief Title: Omega-3 Pufa and Aspirin as Adjunctive Therapy in Treatment of Smoker Patients With Stage Iii Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0710-06/2023
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Diabete Mellitus
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus | interventions — Docosahexaenoic Acids; Aspirin; Doxycycline; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega-3 PUFA and Aspirin (Experimental)
  Interventions: Other: Omega-3 PUFA and Aspirin as adjunctive therapy to (SRP)
- Omega-3 PUFA and Aspirin and doxycycline (Experimental)
  Interventions: Other: Omega-3 PUFA and Aspirin and doxycycline as adjunctive therapy to (SRP)
- Conventional (Active Comparator)
  Interventions: Other: scaling and root planning (SRP)

INTERVENTIONS:
Other: Omega-3 PUFA and Aspirin as adjunctive therapy to (SRP) — fifteen patients will receive ω-3 PUFA + ASA (1g of fish oil/day + 75mg ASA/day for 2 months) after periodontal debridement (TG1)
  Arms: Omega-3 PUFA and Aspirin
Other: Omega-3 PUFA and Aspirin and doxycycline as adjunctive therapy to (SRP) — fifteen patients will receive ω-3 PUFA + ASA (1g of fish oil/day + 75mg ASA/day for 2 months) and oral dosage of doxycycline (100mg every 12 hours on day 1, then 100 mg once daily for 6 days) after periodontal debridement (TG2)
  Arms: Omega-3 PUFA and Aspirin and doxycycline
Other: scaling and root planning (SRP) — fifteen patients will receive periodontal debridement (CG)
  Arms: Conventional

SUMMARY:
Background: Smoking reduces the effect of non-surgical periodontal therapy, a host modulation regimen consisting of omega-3 polyunsaturated fatty acids (ω-3 PUFA) supplementation with low-dose aspirin (ASA) with or without systemic doxycycline has been proposed to improve treatment response.

The Aim of the study is to explore the clinical effects of orally administered omega-3 PUFA and ASA with or without systemic doxycycline with periodontal debridement in treatment of smoker individuals with stage III periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Smoker patients who smoke ≥ 10 cigarettes per day.
* Stages III, Grades C periodontitis with at least one site with PD≥6 and CAL ≥5 mm.

Exclusion Criteria:

* Scaling and root planning in the previous 6 months(that may confound the effect of treatment)
* Antimicrobial therapy in the previous 6 months(that may confound the effect of treatment)
* Chronic systemic diseases that may have an impact on periodontitis progression (diabetes mellitus).
* Systemic diseases that may contraindicate aspirin or doxycycline taking (kidney and liver diseases)
* Allergy to doxycycline
* Long-term usage of medications that may impair periodontal health
* Allergy to fish/seafood

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
change in probing depth | baseline (t0) and at 3 (t1) and 6 months (t2)
  the distance (in millimeters) from the gingival margin to the base of the gingival sulcus or periodontal pocket.
change in clinical attachment level | baseline (t0) and at 3 (t1) and 6 months (t2)
  the distance (in millimeters) from the cemento-enamel junction (CEJ) to the base of the periodontal pocket.

SECONDARY OUTCOMES:
change in gingival index | baseline (t0) and at 3 (t1) and 6 months (t2)
  score 0: Normal gingiva (pink, firm, no bleeding) score 1: Mild inflammation (Slight color change, Slight edema, No bleeding on probing) score 2:Moderate inflammation (Redness, edema, glazing, Bleeding on probing present) score 3: Severe inflammation (Marked redness and edema, Ulceration, Spontaneous bleeding)
change in bleeding on probing | baseline (t0) and at 3 (t1) and 6 months (t2)
  presence of bleeding from the gingival sulcus or periodontal pocket within ~10 seconds after gentle probing.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt